CLINICAL TRIAL: NCT03927326
Title: On Postoperative Analgesic Requirements in Laparoscopic Colorectal Surgery Patients After Exparel Administration Via Transversus Abdominis Plane Block Versus Surgical Infiltration
Brief Title: Postoperative Analgesia in Laparoscopic Abdominal Surgery After Exparel Via TAP or Local Infiltration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Alan Chang, Resident, School of Medicine: Anesthesiology and Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007182
Record Dates: First submitted 2019-04-18; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative; Anesthesia, Local; Anesthesia; Functional; Anesthesia; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Unblinded randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local infiltration (Experimental): Liposomal bupivacaine (266mg) will be directly infiltrated by the surgeon into the surgical laparoscopic wound sites.
  Interventions: Drug: Exparel 266 MG Per 20 ML Injection
- Transversus abdominis plane block (Experimental): Liposomal bupivacaine (266mg) will be used in a ultrasound guided transversus abdominis plane block.
  Interventions: Drug: Exparel 266 MG Per 20 ML Injection

INTERVENTIONS:
Drug: Exparel 266 MG Per 20 ML Injection — Liposomal bupivacaine

SUMMARY:
This study evaluates differences in how administering liposomal bupivacaine via two different methods affects postoperative pain control in laparoscopic abdominal surgery patients. Half the participants will receive liposomal bupivacaine via a transverses abdominis plane block while the other half will receive liposomal bupivacaine via local infiltration.

DETAILED DESCRIPTION:
Liposomal bupivacaine is a newer formulation of a local anesthetic that is commonly used for local infiltration, peripheral nerve blocks, and neuraxial anesthesia. This new formulation allows the effects of bupivacaine to last up to 72 hours as it is slowly released from a liposome. It is FDA approved for local infiltration and has recently been approved for interscalene blocks.

A transversus abdominis plane block is a fascial plane block that is performed routinely for postoperative pain relief for some abdominal incisions. It is performed by placing local anesthetic between the internal oblique and transverses abdominis muscle planes where it will provide analgesia to several dermatomes of the abdomen in hopes of improving postoperative pain relief and reducing postoperative opioid requirement.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic colorectal surgery at UWMC requiring inpatient stay

Exclusion Criteria:

* Patients on chronic pain mediations equaling or exceeding > 25 morphine daily equivalents
* Patients allergic to bupivacaine
* Patients with ASA status IV, V, or VI
* Patients unable to consent
* Patients that are pregnant
* Patients that are incarcerated
* Patients receiving procedures in addition to laparoscopic colorectal procedure
* Patients on systemic anticoagulation precluding them from regional blocks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
24 hour post operative opioid consumption | 24 hours postoperative
  Listed in morphine daily equivalents.

SECONDARY OUTCOMES:
12 hour post operative opioid consumption | 12 hours postoperative
  Listed in morphine daily equivalents
48 hour post operative opioid consumption | 48 hours postoperative
  Listed in morphine daily equivalents
Pain intensity at 12 hours post operative | 12 hours
  Self reported pain intensity by visual analog scale scored 0-10 (0 = no pain; 10 = worst pain imaginable)
Pain intensity at 24 hours post operative | 24 hours
  Self reported pain intensity by visual analog scale scored 0-10 (0 = no pain; 10 = worst pain imaginable)
Hospital length of stay | Until end of hospital stay, typically 3 days
  How long the patient requires their inpatient stay measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Loland, MD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No
We are not planning on making IPD available to other researchers.

REFERENCES:
- [Background] Bergese SD, Ramamoorthy S, Patou G, Bramlett K, Gorfine SR, Candiotti KA. Efficacy profile of liposome bupivacaine, a novel formulation of bupivacaine for postsurgical analgesia. J Pain Res. 2012;5:107-16. doi: 10.2147/JPR.S30861. Epub 2012 May 1. PMID 22570563
- [Background] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Background] Mulligan RP, Morash JG, DeOrio JK, Parekh SG. Liposomal Bupivacaine Versus Continuous Popliteal Sciatic Nerve Block in Total Ankle Arthroplasty. Foot Ankle Int. 2017 Nov;38(11):1222-1228. doi: 10.1177/1071100717722366. Epub 2017 Aug 8. PMID 28786304
- [Background] Sternlicht A, Shapiro M, Robelen G, Vellayappan U, Tuerk IA. Infiltration of liposome bupivacaine into the transversus abdominis plane for postsurgical analgesia in robotic laparoscopic prostatectomy: a pilot study. Local Reg Anesth. 2014 Dec 12;7:69-74. doi: 10.2147/LRA.S64515. eCollection 2014. PMID 25540595
- [Background] Hadzic A, Abikhaled JA, Harmon WJ. Impact of volume expansion on the efficacy and pharmacokinetics of liposome bupivacaine. Local Reg Anesth. 2015 Dec 7;8:105-11. doi: 10.2147/LRA.S88685. eCollection 2015. PMID 26673040
- [Background] Candiotti KA, Sands LR, Lee E, Bergese SD, Harzman AE, Marcet J, Kumar AS, Haas E. Liposome Bupivacaine for Postsurgical Analgesia in Adult Patients Undergoing Laparoscopic Colectomy: Results from Prospective Phase IV Sequential Cohort Studies Assessing Health Economic Outcomes. Curr Ther Res Clin Exp. 2013 Dec 27;76:1-6. doi: 10.1016/j.curtheres.2013.12.001. eCollection 2014 Dec. PMID 25031661
- [Background] Gastevski D. Infiltration of liposome bupivacaine into the transversus abdominis plane for postsurgical pain management in a 39-year-old female undergoing laparoscopic cholecystectomy. Pain Med. 2014 Aug;15(8):1312-5. doi: 10.1111/pme.12356. Epub 2014 Jan 21. PMID 24612211